CLINICAL TRIAL: NCT00321399
Title: SPARC, Including Its Pilot CT Angiographic Study, is a Prospective, Open-label, Multicenter, Sequentially Sampled, Observational Registry to Define the Clinical Value of Stress Perfusion (Stress SPECT, Stress PET), Noninvasive Angiography (CTA) and Combined Perfusion-anatomy (PET/CT) Studies in Patients With Known or Suspected CAD With Respect to Post-test Resource Utilization and Prediction of Cardiac Death and Non-fatal Myocardial Infarction
Brief Title: Study of Perfusion and Anatomy's Role in Coronary Artery (CAD)
Acronym: SPARC
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Marcelo F. Di Carli, MD, FACC, Chief, Division of Nuclear Medicine, Brigham and Women's Hospital
Other Study IDs: SPARC; NCT00575289 (obsolete NCT alias)
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Known CAD, or Intermediate-high Pretest Likelihood for CAD
Keywords: CORONARY ANATOMY; Coronary Artery Disease; SPECT; PET; PET/CT; CTA
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Three main clinical outcomes will be assessed:

1. Post-test resource utilization as assessed by referral rate to catheterization within 90-days of the index study;
2. Incremental prognostic value and risk stratification for predicting cardiac death and myocardial infarction;
3. Cost-effectiveness

To this end, SPARC is organized with two distinct specific objectives with important differences in patient population and endpoints.

Specific Aim 1: To evaluate the impact of stress perfusion imaging with SPECT or PET, CT Angiography, and hybrid PET-CT on post-test resource utilization.

The primary endpoint of specific aim 1 is to compare the impact of combined myocardial perfusion-coronary anatomy data to that of perfusion only [stress SPECT, stress cardiac PET (without CTA)] and anatomy only (CTA alone) on post-test resource utilization, as measured by referral to cardiac catheterization within 90 days of index noninvasive testing, in patients without CAD.

Secondary endpoints:

1. to compare the diagnostic accuracy for detection of epicardial CAD of stress PET and hybrid PET-CT, stress SPECT, and CTA, as defined by coronary angiography;
2. to compare the referral rate to revascularization within 90 days of cardiac catheterization.

Specific Aim 2: To compare the incremental prognostic value and risk stratification of stress perfusion imaging with SPECT or PET, CT coronary angiography, and combined perfusion-anatomy imaging approaches.

The primary endpoint of specific aim 2 is to compare the incremental value of stress perfusion only (stress PET and stress SPECT), coronary anatomy only (CTA data), and combined perfusion-anatomy studies (PET+CTA and SPECT+CTA) over clinical, historical and stress test data for the prediction of cardiac death and nonfatal myocardial infarction.

Secondary endpoints:

1. to compare the incremental value of these noninvasive imaging approaches over clinical, historical and stress test data for the prediction of a composite endpoint including cardiac death, nonfatal myocardial infarction, late (>6 month from index study) referral to revascularization, or late (>6 month from index study) hospitalization for chest pain or heart failure;
2. to compare the incremental value of these noninvasive imaging approaches over clinical, historical and stress test data for the prediction of all cause mortality. In addition, the ability of these modalities -together and separately- to risk stratify patients is a primary goal of specific aim 2.

ELIGIBILITY:
Inclusion Criteria:

* Referred for a clinical stress SPECT, stress PET, CTA or PET-CT study
* Intermediate to high pretest likelihood for CAD (>.25;as defined by ACC/AHA Stable Angina Guidelines) without prior MI/PCI/CABG. These are considered diagnostic patients.

or

* Documented known CAD as defined by prior MI/PCI/CABG
* Provide signed informed consent to participate in the study

Exclusion Criteria:

* Low pretest likelihood for CAD (<=.25; as defined by ACC/AHA Stable Angina Guidelines).
* Major concomitant noncardiac disease or social condition/situation that in the opinion of the investigator will preclude the patient from participation in the study follow-up.
* Concurrent or prior(within last 30 days) participation in other research studies using investigational drugs or devices.
* Presence of a permanent automated internal cardiac defibrillator (AICD)
* Known non-ischemic cardiomyopathy
* Chest pain at rest within 48 hours prior to the index noninvasive imaging test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known coronary artery disease and patients with suspected CAD and an intermediate-High Likelihood of disease
Sampling Method: Non-Probability Sample
Enrollment: 3019 (Actual)
Dates: Start 2006-06; Primary Completion 2010-03 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo F Di Carli, MD FACC, Principal Investigator — Brigham and Women's Hospital; Rory Hachamovitch, MD Msc FACC, Principal Investigator — University of Southern California
Locations (41):
- United States (40):
  - Cardiovascular Associates, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Heart Center, Huntsville, Alabama
  - Scottsdale Medical Imaging, Scottsdale, Arizona
  - Scripps Center for Integrative Medicine, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - Los Angeles Biomedical Research Inst., Torrance, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale - New Haven VA Hospital, New Haven, Connecticut
  - Cardiac Specialists, Trumbull, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Fugua Heart Center - Piedmont Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Sinai Hosptial of Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hosptial, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Minneapolis Heart Inst., Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Holy Name Hospital, Teaneck, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - NYU Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - St. Francis Hospital - The Heart Center, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Meritcare Hospital, Fargo, North Dakota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Tennessee Heart and Vascular Inst., Hendersonville, Tennessee
  - University of Washington Cardiology & Nuclear Medicine, Seattle, Washington
  - Wisconsin Heart Hospital, Milwaukee, Wisconsin
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Hachamovitch R, Nutter B, Hlatky MA, Shaw LJ, Ridner ML, Dorbala S, Beanlands RS, Chow BJ, Branscomb E, Chareonthaitawee P, Weigold WG, Voros S, Abbara S, Yasuda T, Jacobs JE, Lesser J, Berman DS, Thomson LE, Raman S, Heller GV, Schussheim A, Brunken R, Williams KA, Farkas S, Delbeke D, Schoepf UJ, Reichek N, Rabinowitz S, Sigman SR, Patterson R, Corn CR, White R, Kazerooni E, Corbett J, Bokhari S, Machac J, Guarneri E, Borges-Neto S, Millstine JW, Caldwell J, Arrighi J, Hoffmann U, Budoff M, Lima J, Johnson JR, Johnson B, Gaber M, Williams JA, Foster C, Hainer J, Di Carli MF; SPARC Investigators. Patient management after noninvasive cardiac imaging results from SPARC (Study of myocardial perfusion and coronary anatomy imaging roles in coronary artery disease). J Am Coll Cardiol. 2012 Jan 31;59(5):462-74. doi: 10.1016/j.jacc.2011.09.066. PMID 22281249
- [Derived] Hachamovitch R, Johnson JR, Hlatky MA, Cantagallo L, Johnson BH, Coughlan M, Hainer J, Gierbolini J, Di Carli MF; SPARC Investigators. The study of myocardial perfusion and coronary anatomy imaging roles in CAD (SPARC): design, rationale, and baseline patient characteristics of a prospective, multicenter observational registry comparing PET, SPECT, and CTA for resource utilization and clinical outcomes. J Nucl Cardiol. 2009 Nov-Dec;16(6):935-48. doi: 10.1007/s12350-009-9140-7. PMID 19760338